CLINICAL TRIAL: NCT04982666
Title: Assessing the Role of a Whole-Food, Plant-Based (WFPB) Diet in the Treatment of Active Crohn's Disease
Brief Title: Whole-Food, Plant-Based Diet for Active Crohn's Disease
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Difficulties with recruitment and unable to enroll any subjects
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Amanda M. Johnson, Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 21-000714
Record Dates: First submitted 2021-06-03; First posted 2021-07-29 (Actual); Last update posted 2022-05-26 (Actual); Status verified 2022-05

CONDITIONS: Crohn Disease
Keywords: inflammatory bowel disease; diet; crohn disease
MeSH Terms: conditions — Crohn Disease; Inflammatory Bowel Diseases | interventions — Diet, Plant-Based; FODMAP Diet

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Whole-Food, Plant-Based Diet Group (Experimental): Subjects with a known diagnosis of Crohn's disease will follow a whole-food, plant-based diet for a total of 12 weeks
  Interventions: Other: Whole-Food, Plant-Based Diet
- FODMAP Diet (Active Comparator): Subjects with a known diagnosis of Crohn's disease will follow a FODMAP diet for a total of 12 weeks
  Interventions: Other: FODMAP Diet

INTERVENTIONS:
Other: Whole-Food, Plant-Based Diet — This diet is focused on nutritional needs with natural, minimally-processed plant foods.
  Arms: Whole-Food, Plant-Based Diet Group
Other: FODMAP Diet — An elimination diet of fermentable, oligosaccharides, disaccharides, monosaccharides and polyols
  Arms: FODMAP Diet

SUMMARY:
The purpose of this study is to assess the ability of a whole-food, plant-based (WFPB) diet to produce symptomatic remission in Crohn's Disease patients.

DETAILED DESCRIPTION:
The goal of this proposal is to evaluate the efficacy of a whole-food, plant-based (WFPB) diet in the treatment of active Crohn's Disease (CD). Epidemiologic studies suggest that environmental factors, including diet, likely play a role in the pathogenesis and disease course of Inflammatory Bowel Disease (IBD). Evidence also exists to support the idea that dietary practices, such as adherence to a plant-based as opposed to a more "western" diet, can significantly modify the microbiome composition and intestinal barrier function - both of which likely impact the disease course of IBD. The overall hypothesis is that adoption of a WFPB diet will reduce both symptoms and intestinal inflammation in CD patients, as well as increase microbial diversity. Patients will be randomized to receive education on and adopt either WFPB or FODMAP diet, which will be adhered to for a total of 12 weeks. Two primary outcomes which will be assessed are rates of clinical remission based on sCDAI and also reduction in intestinal inflammatory burden based on fecal calprotectin. Several secondary outcomes will also be reviewed to include assessment for alterations in the gut microbiome and intestinal permeability, rates of clinical response based on sCDAI, changes in systemic inflammation based on CRP, and adherence rates to the diet interventions.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older.
* Have the capacity for informed consent.
* Subjects must carry a diagnosis of CD at time of enrollment; the CD diagnosis will be based on clinical impression and documentation of the treating physician.
* Have active symptoms based on sCDAI score of > 175.
* Have active inflammation documented by either: a fecal calprotectin of >150 µg/g; OR high sensitivity C-reactive protein (hs-CRP) >5 mg/L; OR evidence of active inflammation on CT (Computer Tomography) or MR (Magnetic Resonance) enterography, based on discretion of reviewing radiologist; OR documentation of active Crohn's disease on colonoscopy, defined as SES-CD (Simple Endoscopic Score for Crohn's disease) score of 3 or greater.
* Patients may continue their currently prescribed, stable doses of medical therapy during the study duration.
* Ability to have no more than 2 drinks/day for men and 1 drink/day for women.
* Ability and willingness to adhere to one of the study diets.

Exclusion Criteria:

* Hospitalized patients.
* Disease activity score sCDAI > 400
* Already following plant-based diet, FODMAP diet, or other nutritional trials.
* Have recent changes in medical therapy (no start or change in immunomodulator, natalizumab, or vedolizumab within 12 weeks; 5-ASA, anti-TNFα agent, ustekinumab, or tofacitinib within 8 weeks; or corticosteroids within 2 weeks of randomization).
* Have an ostomy or ileoanal pouch.
* Have known luminal stricture or stenosis that would preclude consumption of fresh fruits and vegetables.
* Plans for GI surgery within six weeks of enrollment.
* Pregnant, planning to become pregnant, or breastfeeding.
* Have other conditions such as diabetes or celiac disease that may impact ability to follow study diet.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-04 (Estimated); Primary Completion 2022-06 (Estimated); Study Completion 2022-10 (Estimated)

PRIMARY OUTCOMES:
Change in symptomatic remission | Baseline, week 6, week 12
  Assessed utilizing the short Crohn's Disease Activity Index (sCDAI)
Change in intestinal inflammation | Baseline, week 6, week 12
  Assessed by fecal calprotectin levels. Elevated baseline levels of fecal calprotectin will be defined as >150 µg

SECONDARY OUTCOMES:
Assess the ability of WFPB diet to improve rates of symptomatic response based on sCDAI | Will be evaluated at Visit 3 (week 6) and Visit 4 (week 12) for comparison to baseline.
  Clinical response will be assessed based on changes in sCDAI, with response defined as reduction in sCDAI ≥ 100 as compared to baseline.
Measure the reduction of systemic inflammation based on hsCRP | Will obtain levels at Visit 3 (week 6) and Visit 4 (week 12), for comparison to baseline levels prior to dietary intervention.
  Will be evaluated by comparing changes in high-sensitivity C-reactive protein (hsCRP), with reduction in systemic inflammation defined as normalization in hs-CRP to <5 mg/L.
Assess rates of adherence to diet interventions | This will be administered at Visit 1 (to understand baseline), Visit 3 (week 6), and Visit 4 (week 12).
  Will assess rates of adherence by utilizing Viocare food frequency questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Amanda M Johnson, MD, Principal Investigator — Mayo Clinic

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials